CLINICAL TRIAL: NCT05750121
Title: Effects of E-health Enhanced Motor-cognitive Training on Cognitive Functions, Physical Frailty and Physical Functions of Accident and Emergency Department Discharged Community-dwelling Older Adults With Cognitive Frailty: A Pilot Trial
Brief Title: E-health Enhanced Motor-cognitive Training for AED Discharged Older Adults With Cognitive Frailty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Tung Wah College (Other); Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Dr Daphne Cheung, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HSEARS20220307001
Record Dates: First submitted 2023-01-19; First posted 2023-03-01 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Frailty; Mild Cognitive Impairment
Keywords: Cognitive frailty; Motor-Cognitive Training; Older Adults; Discharged
MeSH Terms: conditions — Frailty; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: 1. Care providers are not included in the study and will not be informed about the group assignment.
  2. An independent administrator will allocate the identifier to the participants and randomise the participants into groups. The administrator will not be involved in the analysis, data collection, outcome assessments, and intervention delivery.
  3. All assessments were conducted by a registered nurse blinded to grouping allocation and will not be involved in intervention training.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): The intervention group will receive home-based motor-cognitive training and usual emergency care.
  Interventions: Behavioral: E-health enhanced motor-cognitive training
- Usual care group (No Intervention): Usual care includes wound care, community nurse service, medications and on-site physiotherapy, occupational therapy, community nurse service, medical social work service, and geriatric nurse follow-up service will be referred when necessary.

INTERVENTIONS:
Behavioral: E-health enhanced motor-cognitive training — The intervention group will implement physical activity (aerobic exercise and resistance training) and cognitive training (CogniFit) intervention with the e-health components (persuasive technology). The intervention period will last for 12 weeks, with three 90 minutes sessions (60 minutes of physical activity and 30 minutes of cognitive training) per week.
  Arms: Treatment group

SUMMARY:
The goal of this pilot randomized controlled trial is to explore the feasibility of e-health enhanced motor-cognitive interventions for discharged community-dwelling older adults with cognitive frailty in the emergency department and to evaluate the effectiveness of the interventions on (1) cognitive functions, (2) physical functions and (3) frailty status.

Participants in the intervention group will receive three-90-minute weekly physical and cognitive training for 12 weeks, facilitated with persuasive technology on smartphones, in addition to the usual care. The control group will receive the usual care. Researchers will explore the feasibility and compare the changes of outcomes between two groups.

DETAILED DESCRIPTION:
Motor-cognitive training effectively reverses and prevents further deterioration of cognitive function, frailty status, and physical function in older adults with cognitive frailty. Recent systematic reviews showed that older adults with cognitive frailty are more likely to develop dementia and have falls than those with frailty alone. The current time-pressured Accident and Emergency Department (AED) setting is challenging for the practitioners to have an intervention to maintain or improve the current physical and cognitive function of these older adults with non-acute complaints and prone to further deteriorate after being discharged from AED. There is a mismatch of services in traditional emergency medicine with the demand of the elderly population. Particular intervention for these older adults is needed. Based on the systematic review and the previous literature, motor-cognitive training is an essential intervention component. Interventions in a home setting can increase flexibility and improve adherence to the intervention. However, the effect on motor-cognitive training in a home setting is unknown. This study aims to explore the feasibility of e-health enhanced motor-cognitive interventions for discharged community-dwelling older adults with cognitive frailty in the emergency department and to evaluate the effectiveness of the interventions on (1) cognitive functions, (2) physical functions and (3) frailty status.

This study is a single-blinded pilot randomised, controlled study. Subjects will be allocated to either the intervention or control group by a 1:1 ratio, where they will receive motor-cognitive training in addition to usual care or usual care only. The program will be targeted older adults aged 60 or above with cognitive frailty and discharged from AED. The intervention lasts for 12 weeks, with three 90 minutes sessions (60 minutes of physical activity and 30 minutes of cognitive training) per week. Trained emergency nurses will provide respective assessments and interventions separately. The primary outcomes are to check the feasibility, including compliance, adherence and adverse effect of the study. Intervention efficacy is the secondary outcome, including physical frailty level, physical performance, and cognitive function. Fried Frailty Index will measure frailty level, physical performance will be measured by Timed-Up-Go Test, handgrip strength, gait speed, chair stand test, arm curl test and Physical Activity Scale for the Elderly. Montreal cognitive assessment (MoCA), Fuld object-memory evaluation (FOME), trail making test (TMT) will be used to measure the cognitive functions. Secondary outcome indicators included. Data will be collected in two-time points, baseline and post-intervention Findings of the study can help in improving the actual research and providing evidence for implementing motor-cognitive training for AED-discharged older adults with cognitive frailty.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years old or above;
* discharged from the AED;
* Cantonese speaking;
* have a smartphone and have experience in using the smartphone for at least six months;
* with cognitive frailty, the coexistence of mild cognitive impairment (MCI) and physical frailty, without being diagnosed as dementia.

Exclusion Criteria:

* unable to make consent,
* unable to communicate due to language barrier or visual impairment or uncorrectable hearing impairment,
* old aged home residents,
* already participated in other interventional studies,
* participate in any geriatric program and training, or
* impaired mobility

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2024-01-29 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | At baseline
  One of the feasibility outcomes. It is the overall recruitment rate, which will be calculated by dividing the number of recruited and randomized, by the total invited eligible potential participants. It will range from 0 to 100%.
Retention rate | At the 12th - 14th week (post-intervention)
  One of the feasibility outcomes. It is calculated by dividing the number of randomised participants retained and assessed with valid primary outcome data at the end of the project, by the recruited participants. It will range from 0 to 100%.
Adverse events | Continuous monitoring throughout the 12 weeks of intervention
  A feasibility indicators, which is defined as an undesired effect of the intervention. Any adverse events reported by the participants will be documented and reported.

SECONDARY OUTCOMES:
Global cognition | At baseline, and the 12th - 14th week (post intervention)
  It will be assessed with the Hong Kong version Montreal of Cognitive Assessment. The total score of the instrument ranges from 0 - 30. Higher score indicates better cognitive functions.
Memory | At baseline, and the 12th - 14th week (post intervention)
  It will be measured with Fuld Object Memory Evaluation. It consists of three subscores, namely the total storage, total retrieval and delayed recall with the highest possible scores of 50, 50, and 10 respectively. Higher the scores indicate better cognitive functions.
Visual attention and task switching | At baseline, and the 12th - 14th week (post intervention)
  It will be measured with the Trail Making Test (TMT), which consists of two parts: TMT-A and TMT-B. Shorter the time used indicates better cognitive functions.
Mobility | At baseline, and the 12th - 14th week (post intervention)
  It will be measured with the Time-up-and-Go test. It represents the total time needed for the participants to stand and walk for 3 meters, turn around and walk back to the chair and sit down. Shorter the time used indicates better monility.
Gait speed | At baseline, and the 12th - 14th week (post intervention)
  The time used for the 6-meter walk, shorter the time used indicates better gait speed.
Leg strength and endurance | At baseline, and the 12th - 14th week (post intervention)
  It will be assessed with the Chair Stand Test. The participants will be required to stand up repeatedly from a chair for 30 seconds. The higher number of stands a person can complete in 30 seconds, indicates a better leg strength and endurance.
Physical activity | At baseline, and the 12th - 14th week (post intervention)
  It will be measured with the Physical Activity Scale for the Elderly, which quantify the amount of daily physical activity. The total score ranges from 0 to 793, with a higher score indicates a larger amount of physical activity.
Hand-grip strength | At baseline, and the 12th - 14th week (post intervention)
  It will be measured with a handgrip dyanometer.
Strength of upper extremities | At baseline, and the 12th - 14th week (post intervention)
  It will be measured with the Arm-Curl Test. The number of bicep curls in 30 seconds while holding a hand weight.
Actigraph data | Throughout the 12 weeks intervention period.
  Data will be collected with a wrist worn Actigraph GT3X+ device.
Frailty status | At baseline, and the 12th - 14th week (post intervention)
  The Fried Frailty Index will be used to measure the frailty status. The total score ranges from 0 to five. Higher score indicates a higher frailty level. Score 0, 1-2, and 3-5 correspond to robust, pre-frail, and frail respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing, The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided